CLINICAL TRIAL: NCT07295938
Title: A Study to Assess the Traditional Chinese Medicine as Adjunctive Therapy to Improve Cure Rates During the Continuation Phase in Mycobacterium Abscessus Pulmonary Disease
Brief Title: TCM as an Adjuvant Treatment in Mycobacterium Abscessus Pulmonary Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other); Anhui Chest Hospital (Other); Guangzhou Chest Hospital. (Unknown); Jiangxi Chest Hospital (Unknown); Beijing Chest Hospital (Other); China-Japan Friendship Hospital (Other); Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhenhui Lu, chief physician, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024LCSY166
Record Dates: First submitted 2025-11-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Mycobacterium Abscessus Pulmonary Disease
Keywords: Mycobacterium abscessus Pulmonary Disease; Continuation Phase; TCM

STUDY DESIGN:
Intervention Model Description: All participants in the treatment group received the recommended treatment regimen according to guidelines, supplemented with Chinese herbs, upon study entry. In contrast, the control group received a placebo consisting of a 1/20 dose of Chinese herbs.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a Double-blind Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Group-I (Experimental): 104 participants with persistently positive bacterial cultures during the continuation phase received Chinese herbal therapy in addition to the guideline-recommended regimen, with the primary endpoint being the cure rates at 52 weeks.
  Interventions: Drug: Chinese herbs-I
- Control Group-I (Placebo Comparator): 104 participants with persistently positive bacterial cultures during the continuation phase received a placebo comprising a 1/20 dose of Chinese herbs in addition to the guideline-recommended regimen, with the primary endpoint being the cure rates at 52 weeks.
  Interventions: Drug: Chinese herbs-I placebo
- Treatment Group-II (Experimental): 72 participants with negative bacterial cultures during the continuation phase received Chinese herbal therapy in addition to the guideline-recommended regimen, with the primary endpoint being the relapse or reinfection rates at 52 weeks.
  Interventions: Drug: Chinese herbs-II
- Control Group-II (Placebo Comparator): 72 participants with negative bacterial cultures during the continuation phase received a placebo comprising a 1/20 dose of Chinese herbs in addition to the guideline-recommended regimen, with the primary endpoint being the relapse or reinfection rates at 52 weeks.
  Interventions: Drug: Chinese herbs-II placebo

INTERVENTIONS:
Drug: Chinese herbs-I — This is an empirical traditional Chinese medicine compound used in the treatment of Mycobacterium abscessus pulmonary disease for a long time
  Arms: Treatment Group-I
Drug: Chinese herbs-I placebo — Chinese herbs-I placebo
  Arms: Control Group-I
Drug: Chinese herbs-II — This is an empirical traditional Chinese medicine compound used in the treatment of Mycobacterium abscessus pulmonary disease during the continuation phase for a long time
  Arms: Treatment Group-II
Drug: Chinese herbs-II placebo — Chinese herbs-II placebo
  Arms: Control Group-II

SUMMARY:
Chinese herbs can facilitate sputum culture conversion, promote lesion absorption, and enhance clinical symptoms and quality of life for patients with Mycobacterium abscessus pulmonary disease (MAB-PD). The investigators aimed to evaluate the efficacy of Chinese herbs as adjunct therapy to improve cure rates or reduce recurrence rates during the continuation phase of MAB-PD treatment.

DETAILED DESCRIPTION:
Mycobacterium abscessus pulmonary disease (MAB-PD) is a significant form of non-tuberculous mycobacterial lung infection that clinically presents with symptoms such as cough, sputum production, hemoptysis, low-grade fever, and chest tightness. Current guidelines recommend treatment regimens that are divided into initial and continuation phases. The initial phase involves combination therapy with at least three antibiotics, which can be administered intravenously or orally. In contrast, the continuation phase requires the use of oral or inhaled antibiotics. Guidelines suggest continuing treatment for 12 months after sputum culture negativity, although standard protocols indicate only a 35% cure rate with up to a 40% post-treatment relapse rate. Research has shown that traditional Chinese herbal formulas have broad immunomodulatory effects, which promote sputum culture conversion, lesion absorption, and improvement in clinical symptoms and quality of life for patients with MAB-PD. This study will enroll patients with MAB-PD who have completed initial treatment and will be divided into two independent randomized controlled trials (RCTs) based on sputum M.abscessus culture results. RCT-1 will include patients with persistently positive bacterial cultures receiving Chinese herbal therapy supplemented with the guideline-recommended regimen, with primary endpoints being 52-week cure rates. RCT-2 will include patients with negative bacterial cultures receiving Chinese herbal therapy supplemented with the guideline-recommended regimen, with primary endpoints being 52-week rates of relapse or reinfection. Patients will receive complimentary Chinese herbal medicine. All participants will undergo sputum or bronchoalveolar lavage fluid bacteriological testing, chest imaging, pulmonary function tests, a 6-minute walk test, SF-36, QOL-B, SGRQ, and HADS scales. Additionally, exploratory studies will collect sputum, bronchoalveolar lavage fluid, blood, and stool samples to identify the comprehensive immune profile of MAB-PD and evaluate the intervention advantages of traditional Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with Mycobacterium abscessus pulmonary disease;
* Patients have completed the initial phase of treatment as recommended by the guidelines;
* Patients who have given written informed consent
* One week prior to enrollment, organ function levels must meet the following criteria: a. Hemoglobin ≥60g/L; b. Neutrophil count ≥0.5×10^9/L; c. Platelet count ≥60×10^9/L; d. Serum total bilirubin ≤3 times the upper limit of normal; e. Aspartate aminotransferase ≤3 times the upper limit of normal; f. Alanine aminotransferase ≤3 times the upper limit of normal; g. Creatinine level below 2 times the upper limit of normal or creatinine clearance ≥60mL/min; h. Urea nitrogen ≤200mg/L; i. Urinary protein <++, with ≥500mg total protein in 24-hour urine if protein is present; j. Blood glucose: within normal range and/or stable blood glucose control in diabetic patients; k. Cardiac function: no history of myocardial infarction within 6 months; no unstable angina; no severe arrhythmia.

Exclusion Criteria:

* Patients with a drug allergy to the investigational medication;
* Patients infected with two or more non-tuberculous mycobacteria, or those with active pulmonary tuberculosis;
* Patients with a prior history of pulmonary parenchymal organ transplantation;
* Patients with severe conditions such as congenital or acquired immunodeficiency disorders, active malignant tumors (primary or metastatic), or any malignancies requiring chemotherapy or radiotherapy during screening or study;
* Patients undergoing dialysis;
* Patients with radiation pneumonitis requiring corticosteroid or immunoglobulin pulse therapy, or clinically proven active interstitial lung disease, uncontrolled massive pleural effusion, or pericardial effusion;
* Unstable systemic comorbidities (hypertensive crisis, unstable angina, congestive heart failure, myocardial infarction within the past 6 months, severe psychiatric disorders requiring medication, severe hepatic or renal dysfunction, neuropsychiatric conditions such as Alzheimer's disease);
* Patients with intestinal dysfunction or malabsorption syndrome;
* Pregnant or breastfeeding women;
* Patients receiving other investigational drugs within 4 weeks prior to first exposure to the study drug;
* Concurrent enrollment in another clinical trial, except for observational (non-interventional) studies or follow-up visits in interventional trials;
* Physical examinations or clinical tests that the investigator deems potentially interfering with results or increasing treatment-related complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate | At the end of 52 weeks of treatment
  Measured the change from the Baseline to the end of treatment. The sputum MAB culture was negative on three consecutive occasions, with at least a one-month interval between each, and there were no subsequent positive results.
Relapse or reinfection rates | At the end of 52 weeks of treatment
  Bacterial relapse is defined as the occurrence of at least two cultures and/or molecular biology tests identifying the same pathogenic M. abscessus strain as the initial infection after completing anti-M. abscessus treatment. When necessary, genotyping techniques may be employed to differentiate between relapse and reinfection. Reinfection refers to the emergence of different pathogenic strains or species in at least two positive cultures following the initiation of treatment.

SECONDARY OUTCOMES:
Time to sputum culture conversion | From baseline to 52 weeks post-treatment completion
  Measured the change from Baseline to the end of treatment
Absorption rate of lung lesions | Baseline, 26 weeks and 52 weeks
  The lung lesion absorption rate is assessed via chest imaging to evaluate changes in pulmonary infection lesions compared to the baseline at 26 and 52 weeks after enrollment. Patients with more than half of their lesions absorbed are classified as showing significant absorption; those with less than half absorption are considered to have absorption; those with no changes are deemed to show no change; and those with enlarged lesions or new lesions are regarded as demonstrating deterioration. The determination of the lung lesion absorption rate is made by professional radiology experts.
Rate of closure of lung cavities | Baseline, 26 weeks and 52 weeks
  The lung cavity closure rate is assessed through chest imaging to evaluate changes in lung cavities compared to the baseline at 26 and 52 weeks after enrollment. The clinical criteria for CT changes were as follows: Regarding changes in cavity size, scar healing, block healing, or disappearance were defined as closure. A reduction in cavity size by 1/2 or more was defined as reduction, a reduction in cavity diameter by less than 1/2 was classified as no change, and an increase in the cavity diameter by 1/2 or more was defined as increase.
  The determination of the lung lesion absorption rate is made by professional radiology experts.
Pulmonary function tests | Baseline, 26 weeks and 52 weeks
  Assess the patient's pulmonary function, specifically the changes in FEV1 (L), before treatment, as well as at 26 weeks and 52 weeks post-treatment
6 minute walking test | Baseline, 12 weeks, 26 weeks, 40 weeks and 52 weeks
  Measured the change from Baseline to the end of treatment
36 - item Short Form (SF - 36) | Baseline, 12 weeks, 26 weeks, 40 weeks and 52 weeks
  The 36 - item Short Form (SF - 36) consists of 8 domains, namely physical functioning, role-physical, bodily pain, general health perceptions, vitality, social functioning, role-emotional, and mental health. The SF - 36 scale ranges from 0 to 100 points, where higher scores signify better outcomes. The change from baseline to the end of treatment was measured at the indicated time.
Quality of Life Questionnaire for Bronchiectasis (QoL-B) | Baseline, 12 weeks, 26 weeks, 40 weeks and 52 weeks
  The Quality of Life Questionnaire for Bronchiectasis (QoL-B) encompasses eight dimensions: physical function, role function, vitality, emotion, social function, treatment effect, health perception, and respiratory symptoms. Each dimension is scored on a scale ranging from 0 to 100, where higher scores signify a better quality of life. The change from baseline to the end of treatment was measured at the indicated time.
Saint George's respiratory questionnaire (SGRQ) | Baseline, 12 weeks, 26 weeks, 40 weeks and 52 weeks
  The Saint George's Respiratory Questionnaire (SGRQ) scale comprises 50 questions, which assess three aspects: symptoms, activity, and disease impact. The calculation method is a weighted - average algorithm. The score of each item ranges from 0 to 100. The higher the score, the poorer the quality of life; the lower the score, the better the quality of life. The change from the baseline to the end of treatment was measured at the indicated time.
Hospital Anxiety and Depression Scale (HADS) | Baseline, 12 weeks, 26 weeks, 40 weeks and 52 weeks
  The HADS scale is employed to evaluate patients' anxiety and depression, with a total score ranging from 0 to 42 points. The anxiety sub - scale ranges from 0 to 21 points, and the depression sub - scale also ranges from 0 to 21 points. Higher scores signify a greater risk of anxiety or depression. The change from the baseline to the end of treatment was measured at the specified time.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenhui Lu, Study Chair — Longhua Hospital
Locations (8):
- China (8):
  - Beijing Chest Hospital Affiliated to Capital Medical University, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Guangzhou Municipal Hospital of Chest Medicine, Guangdong
  - Anhui Provincial Chest Hospital, Hefei
  - Jiangxi Chest Hospital, Nanchang
  - Fudan University Affiliated Huashan Hospital, Shanghai
  - Longhua Hospital Affiliated Shanghai University of TCM, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai